CLINICAL TRIAL: NCT03336281
Title: Prospective, Multicenter, Non-interventional Study to Characterize Profile of Patient With Psoriatic Arthritis Depending on Whether Their Disease is Managed by a Dermatologist or by a Rheumatologist, and Starting Ustekinumab
Brief Title: A Study to Characterize Profile of Participant With Psoriatic Arthritis Depending on Whether Their Disease is Managed by a Dermatologist or by a Rheumatologist, and Starting Ustekinumab
Acronym: PROUST
Status: Completed | Type: Observational
Sponsor: Janssen Cilag S.A.S. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108343; CNTO1275PSO4058 (Other: Janssen Cilag S.A.S., France)
Record Dates: First submitted 2017-11-03; First posted 2017-11-08 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Psoriatic Arthritis: Dermatologist Cohort: Participants who will receive ustekinumab (as a first or second line of biologic disease modifying anti-rheumatic drug [bDMARD] therapy) along with other co-medications as per clinical dematologist's discretion will be observed in this study. Ustekinumab will not be provided by the sponsor. The treatment by ustekinumab must have been decided by the physician prior to the decision to include the participant in the study. Only data available from a participant's source medical records will be collected. Additionally investigators will be asked to obtain (or record where available) Patient-Reported Outcome (PRO) data from participants participating in this study.
  Interventions: Drug: Ustekinumab
- Participants with Psoriatic Arthritis: Rheumatologist Cohort: Participants who will receive ustekinumab (as a first or second line of bDMARD therapy) along with other co-medications as per clinical rheumatologist's discretion will be observed in this study. Ustekinumab will not be provided by the sponsor. The treatment by ustekinumab must have been decided by the physician prior to the decision to include the participant in the study. Only data available from a participant's source medical records will be collected. Additionally investigators will be asked to obtain (or record where available) PRO data from participants participating in this study.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — All participants will receive ustekinumab at study entry. Ustekinumab will not be provided by the sponsor. The treatment decision must have been taken by the investigator prior to, and independently of the participant's inclusion into the study following the standard clinical practice. Only data available from a participant's source medical records will be collected.

SUMMARY:
The primary purpose of this study is to describe the Psoriatic Arthritis (PsA) participant profiles depending on whether their disease is managed by a dermatologist or by a rheumatologist in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Participant with a confirmed diagnosis of Psoriatic Arthritis (PsA) according to the dermatological and/or rheumatologic routine practice, using different diagnosis tools, example, the Classification criteria for Psoriatic Arthritis (CASPAR), or others
* Participant must be starting ustekinumab for PsA according to the local labelling, as a first (biological naïve participant), or second line (biological experienced participants) of bDMARD therapy: First line bDMARD therapy: The first line therapy includes all bio-naïve participants who start their ustekinumab as their first biologic treatment at the study start (within a maximum 1-month window after the baseline visit); Second line bDMARD therapy: The second line therapy includes participants who initiated ustekinumab as their second biologic therapy at the study start (within a maximum 1-month window after the baseline visit)
* Participant for which the ustekinumab treatment has been decided by the investigator prior to and independently of the participant's inclusion into the study
* Participant for which the first administration of the ustekinumab treatment will occur within the 4-week period from inclusion assessment
* Participant has signed an informed consent form

Exclusion Criteria:

* Participant starting ustekinumab as a third or further line of bDMARD therapy
* Already ustekinumab-experienced participants
* Participant has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within at least 30 days before the start of the study or more according to the half-life of the investigational drug
* Participant has refused to participate in the study or unable to give his consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a confirmed diagnosis of Psoriatic Arthritis (PsA) according to the clinical practice and for which a treatment with ustekinumab is indicated as a first (biological-naïve participants) or a second line (biological-experienced participants) of biological disease-modifying antirheumatic drugs (bDMARD) for PsA / psoriasis (PsO) will be observed depending on whether their disease is managed by a dermatologist or by a rheumatologist in routine practice.
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Swelling of Joints at Baseline | Baseline (Week 0)
  Participants with swollen 28-joints or 66/68-joints counts according to the practices will be evaluated.
Number of Participants With Swelling of Joints at Week 16 | Week 16
  Participants with swollen 28-joints or 66/68-joints counts according to the practice will be evaluated.
Number of Participants With Swelling of Joints at Week 28 | Week 28
  Participants with swollen 28-joints or 66/68-joints counts according to the practice will be evaluated.
Number of Participants With Tenderness of Joints at Baseline | Baseline (Week 0)
  Participants with tender 28-joints or 66/68-joints counts according to the practice will be evaluated.
Number of Participants With Tenderness of Joints at Week 16 | Week 16
  Participants with tender 28-joints or 66/68-joints counts according to the practice will be evaluated.
Number of Participants With Tenderness of Joints at Week 28 | Week 28
  Participants with tender 28-joints or 66/68-joints counts according to the practice will be evaluated.
Change From Baseline in Disease Activity Score in 28 Joints (DAS28) at Week 16 | Baseline and Week 16
  The DAS28 score is a measure of the participant's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], participant's global assessment of disease activity [visual analog scale: 0 = no disease activity to 100 = maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 (best) to approximately 10 (worst). Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from baseline indicated improvement.
Change From Baseline in Disease Activity Score in 28 Joints (DAS28) at Week 28 | Baseline and Week 28
  The DAS28 score is a measure of the participant's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], participant's global assessment of disease activity [visual analog scale: 0 = no disease activity to 100 = maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 (best) to approximately 10 (worst). Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from baseline indicated improvement.
Percentage of Participants Achieving European League Against Rheumatism (EULAR) Good Response at Baseline | Baseline (Week 0)
  Clinical response will be assessed according to EULAR categorical DAS28 response criteria. DAS28 score: participant's disease activity calculated using TJC28, SJC28, PGH [VAS: 0=no disease activity to 100=maximum disease activity] and ESR. Total possible score = 0-10, higher scores represented higher disease activity. EULAR Good response: DAS28 less than or equal to (<=) 3.2 or a change from baseline less than (<) -1.2.
Percentage of Participants Achieving EULAR Good Response at Week 16 | Week 16
  Clinical response will be assessed according to EULAR categorical DAS28 response criteria. DAS28 score: participant's disease activity calculated using TJC28, SJC28, PGH [VAS: 0=no disease activity to 100=maximum disease activity] and ESR. Total possible score = 0-10, higher scores represented higher disease activity. EULAR Good response: DAS28 <= 3.2 or a change from baseline < -1.2.
Percentage of Participants Achieving EULAR Good Response at Week 28 | Week 28
  Clinical response will be assessed according to EULAR categorical DAS28 response criteria. DAS28 score: participant's disease activity calculated using TJC28, SJC28, PGH [VAS: 0=no disease activity to 100=maximum disease activity] and ESR. Total possible score = 0-10, higher scores represented higher disease activity. EULAR Good response: DAS28 <= 3.2 or a change from baseline < -1.2.
Percentage of Participants Achieving Minimal Disease Activity (MDA) at Baseline | Baseline (Week 0)
  The MDA is a state of disease activity deemed a useful target of treatment by both the participant and physician. The percentage of participants achieving MDA will be determined based on participants fulfilling 5 of the following 7 criteria must be met: Tender joint count <= 1; Swollen joint count <= 1; psoriasis area and severity index (PASI) <= 1 or BSA <= 3; Participant pain VAS <= 15; Participant global activity VAS <= 20; Health Assessment Questionnaire (HAQ) <= 0.5; Tender enthesial points <= 1.
Percentage of Participants Achieving MDA at Week 16 | Week 16
  The MDA is a state of disease activity deemed a useful target of treatment by both the participant and physician. The percentage of participants achieving MDA will be determined based on participants fulfilling 5 of the following 7 criteria must be met: Tender joint count <= 1; Swollen joint count <= 1; PASI <= 1 or BSA <= 3; Participant pain VAS <= 15; Participant global activity VAS <= 20; HAQ <= 0.5; Tender enthesial points <= 1.
Percentage of Participants Achieving MDA at Week 28 | Week 28
  The MDA is a state of disease activity deemed a useful target of treatment by both the participant and physician. The percentage of participants achieving MDA will be determined based on participants fulfilling 5 of the following 7 criteria must be met: Tender joint count <= 1; Swollen joint count <= 1; PASI <= 1 or BSA <= 3; Participant pain VAS <= 15; Participant global activity VAS <= 20; HAQ <= 0.5; Tender enthesial points <= 1.
Change from Baseline in Physician's Global Assessment of Disease Activity - Psoriatic Arthritis (PGA-PsA) Visual Analogue Scale (VAS) Scores at Week 16 | Baseline and Week 16
  Physician's Global Assessment of Disease Activity (PGA-PsA) will be measured using a visual analogue scale with scores ranging from 0 to 100 (higher scores indicate worse disease activity).
Change from Baseline in PGA-PsA VAS Scores at Week 28 | Baseline and Week 28
  Physician's Global Assessment of Disease Activity (PGA) will be measured using a visual analogue scale with scores ranging from 0 to 100 (higher scores indicate worse disease activity).
Change from Baseline in Patient's Global Assessment (PtGA-PsA) VAS Scores at Week 16 | Baseline and Week 16
  The PtGA by VAS measuring the overall way the disease affects the participants at a point in time. The score will be recorded as a single vertical mark on a 100 millimeter (mm) visual analogic scale (VAS), with 0 representing the lowest level of disease activity and 100 representing the highest.
Change from Baseline in PtGA-PsA VAS Scores at Week 28 | Baseline and Week 28
  The PtGA by VAS measuring the overall way the disease affects the participants at a point in time. The score will be recorded as a single vertical mark on a 100 millimeter (mm) visual analogic scale (VAS), with 0 representing the lowest level of disease activity and 100 representing the highest.
Participant's Pain VAS Scores at Baseline | Baseline (Week 0)
  The score will be recorded as a single vertical mark placed by participant on a 100 mm visual analogic scale (VAS), with 0 representing the no pain of and 100 representing the highest pain as severe as can be imagined. The distance from the mark will be recorded.
Participant's Pain VAS Scores at Week 16 | Week 16
  The score will be recorded as a single vertical mark placed by participant on a 100 mm visual analogic scale (VAS), with 0 representing the no pain of and 100 representing the highest pain as severe as can be imagined. The distance from the mark will be recorded.
Participant's Pain VAS Scores at Week 28 | Week 28
  The score will be recorded as a single vertical mark placed by participant on a 100 mm visual analogic scale (VAS), with 0 representing the no pain and 100 representing the highest pain as severe as can be imagined. The distance from the mark will be recorded.
Percentage of Participants With Dactylitis at Baseline | Baseline (Week 0)
  Percentage of participants with dactylitis will be evaluated.
Percentage of Participants With Dactylitis at Week 16 | Week 16
  Percentage of participants with dactylitis will be evaluated.
Percentage of Participants With Dactylitis at Week 28 | Week 28
  Percentage of participants with dactylitis will be evaluated.
Change from Baseline in Dactylitis Count at Week 16 | Baseline and Week 16
  The change from baseline in total number of digits of the hands and feet (that is, 0 to 20) with dactylitis will be evaluated.
Change from Baseline in Dactylitis Count at Week 28 | Baseline and Week 28
  The change from baseline in total number of digits of the hands and feet (that is, 0 to 20) with dactylitis will be evaluated.
Percentage of Participants With Dactylitis Complete Resolution at Baseline | Baseline (Week 0)
  Percentage of participants with complete resolution of dactylitis in hands and feet will be evaluated.
Percentage of Participants With Dactylitis Complete Resolution at Week 16 | Week 16
  Percentage of participants with complete resolution of dactylitis in hands and feet will be evaluated.
Percentage of Participants With Dactylitis Complete Resolution at Week 28 | Week 28
  Percentage of participants with complete resolution of dactylitis in hands and feet will be evaluated.
Percentage of Participants With Enthesitis at Baseline | Baseline (Week 0)
  Percentage of participants with enthesitis will be evaluated.
Percentage of Participants With Enthesitis at Week 16 | Week 16
  Percentage of participants with enthesitis will be evaluated.
Percentage of Participants With Enthesitis at Week 28 | Week 28
  Percentage of participants with enthesitis will be evaluated.
Change from Baseline in Enthesitis Score at Week 16 | Baseline and Week 16
  Enthesitis will be documented using the Leeds Enthesitis Index (LEI). The LEI evaluates the presence or absence of pain by applying local pressure to lateral epicondyle (left and right), medial femoral condyle (left and right), and Achilles tendon insertion (left and right). LEI Enthesitis Index scores ranging from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness).
Change from Baseline in Enthesitis Score at Week 28 | Baseline and Week 28
  Enthesitis will be documented using the Leeds Enthesitis Index (LEI). The LEI evaluates the presence or absence of pain by applying local pressure to lateral epicondyle (left and right), medial femoral condyle (left and right), and Achilles tendon insertion (left and right). LEI Enthesitis Index scores ranging from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness).
Percentage of Participants With Enthesitis Complete Resolution at Week 16 | Week 16
  Percentage of participants with complete resolution from enthesitis will be evaluated.
Percentage of Participants With Enthesitis Complete Resolution at Week 28 | Week 28
  Percentage of participants with complete resolution from enthesitis will be evaluated.
Change From Baseline in Erythrocytic Sedimentation Rate (ESR) at Week 16 | Baseline and Week 16
  ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 millimeter per hour (mm/hr). A higher rate is consistent with inflammation.
Change From Baseline in ESR at Week 28 | Baseline and Week 28
  ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 millimeter per hour (mm/hr). A higher rate is consistent with inflammation.
Change From Baseline in C-Reactive Protein (CRP) at Week 16 | Baseline and Week 16
  The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Change From Baseline in CRP at Week 28 | Baseline and Week 28
  The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Percentage of Participants With Psoriatic Arthritis (PsA) Extra-articular Manifestations at Baseline | Baseline (Week 0)
  Percentage of participants with PsA extraarticular manifestations will be assessed. Extra-articular manifestations are symptoms and diseases that occur in parts of the body other than joints. These included the presence of enthesitis (inflammation of ligaments and/or tendons at the site of insertion into bones), uveitis (inflammation of the middle layer of the eye), psoriasis (a skin condition that causes itchy or sore patches of thick, red skin with silvery scales), and Inflammatory bowel disease (Crohn's disease or ulcerative colitis).
Percentage of Participants With PsA Extra-articular Manifestations at Week 16 | Week 16
  Percentage of participants with PsA extraarticular manifestations will be assessed. Extra-articular manifestations are symptoms and diseases that occur in parts of the body other than joints. These included the presence of enthesitis (inflammation of ligaments and/or tendons at the site of insertion into bones), uveitis (inflammation of the middle layer of the eye), psoriasis (a skin condition that causes itchy or sore patches of thick, red skin with silvery scales), and Inflammatory bowel disease (Crohn's disease or ulcerative colitis).
Percentage of Participants With PsA Extra-articular Manifestations at Week 28 | Week 28
  Percentage of participants with PsA extraarticular manifestations will be assessed. Extra-articular manifestations are symptoms and diseases that occur in parts of the body other than joints. These included the presence of enthesitis (inflammation of ligaments and/or tendons at the site of insertion into bones), uveitis (inflammation of the middle layer of the eye), psoriasis (a skin condition that causes itchy or sore patches of thick, red skin with silvery scales), and Inflammatory bowel disease (Crohn's disease or ulcerative colitis).
Percentage of Participants With Body Surface Area (BSA) Psoriasis (PsO) Skin Involvement at Baseline | Baseline (Week 0)
  Psoriasis skin involvement will be documented using categories: <3 percent (%), 3% to 10%, and >10% of BSA. The typical method to assess BSA is to consider the surface area of the participant's handprint (palm and fingers) as representing 1% of the body's surface area.
Percentage of Participants With BSA PsO Skin Involvement at Week 16 | Week 16
  Psoriasis skin involvement will be documented using categories: <3 percent (%), 3% to 10%, and >10% of BSA. The typical method to assess BSA is to consider the surface area of the participant's handprint (palm and fingers) as representing 1% of the body's surface area.
Percentage of Participants With BSA PsO Skin Involvement at Week 28 | Week 28
  Psoriasis skin involvement will be documented using categories: <3 percent (%), 3% to 10%, and >10% of BSA. The typical method to assess BSA is to consider the surface area of the participant's handprint (palm and fingers) as representing 1% of the body's surface area.
Change From Baseline in Nail Involvement Scores at Week 16 | Baseline and Week 16
  Nail involvement will be evaluated by recording the total number of nails of the hands and feet (that is, 0 to 20) with PsA involvement.
Change From Baseline in Nail Involvement Scores at Week 28 | Baseline and Week 28
  Nail involvement will be evaluated by recording the total number of nails of the hands and feet (that is, 0 to 20) with PsA involvement.
Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Week 16 | Baseline and Week 16
  The Stanford Health Assessment Questionnaire Disability Index (HAQ-DI) is a participant completed questionnaire specific for rheumatoid arthritis, consisting of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. There are 4 possible responses for each question: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty and 3=unable to do. The score for each of the domains is the highest (worst) score in each domain. A participant must have a domain score for at least 6 of 8 domains to calculate a valid HAQ-DI score which is the sum of domain scores, divided by the number of domains that have a score for a total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from baseline indicated improvement.
Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Week 28 | Baseline and Week 28
  The Stanford Health Assessment Questionnaire Disability Index (HAQ-DI) is a participant completed questionnaire specific for rheumatoid arthritis, consisting of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. There are 4 possible responses for each question: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty and 3=unable to do. The score for each of the domains is the highest (worst) score in each domain. A participant must have a domain score for at least 6 of 8 domains to calculate a valid HAQ-DI score which is the sum of domain scores, divided by the number of domains that have a score for a total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from baseline indicated improvement.
Percentage of Participants Achieving HAQ-DI Response at Baseline | Baseline (Week 0)
  Percentage of participants achieving HAQ-DI response that is change of greater than (>) 0.3 will be evaluated.
Percentage of Participants Achieving HAQ-DI Response | Week 16
  Percentage of participants achieving HAQ-DI response that is change of > 0.3 will be evaluated.
Percentage of Participants Achieving HAQ-DI Response at Week 28 | Week 28
  Percentage of participants achieving HAQ-DI response that is change of > 0.3 will be evaluated.
Change From Baseline in Psoriatic Arthritis Impact of Disease-12 (PsAID-12) Questionnaire Scores at Week 16 | Baseline and Week 16
  The PsAID-12 is a validated, self-administered questionnaire developed by EULAR for use in clinical practice that assesses the impact of PsA on participants' lives. It consists of 12 questions, each answered using a numerical rating scale. Questions related to pain, skin problems, work and/or leisure activities, discomfort, embarrassment and/or shame, social participation, and anger, fear, and uncertainty; and depression are scored from 0 (none) to 10 (extreme), functional capacity and sleep disturbance are scored from 0 (no difficulty) and 10 (extreme difficulty) and coping is scored from 0 (very well) 10 (very poorly).
Change From Baseline in PsAID-12 Questionnaire Scores at Week 28 | Baseline and Week 28
  The PsAID-12 is a validated, self-administered questionnaire developed by EULAR for use in clinical practice that assesses the impact of PsA on participants' lives. It consists of 12 questions, each answered using a numerical rating scale. Questions related to pain, skin problems, work and/or leisure activities, discomfort, embarrassment and/or shame, social participation, and anger, fear, and uncertainty; and depression are scored from 0 (none) to 10 (extreme), functional capacity and sleep disturbance are scored from 0 (no difficulty) and 10 (extreme difficulty) and coping is scored from 0 (very well) 10 (very poorly).
Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score at Week 16 | Baseline and Week 16
  The BASDAI is used to measure the ankylosing spondylitis (AS) disease severity. It consists of 6 questions: fatigue, spinal pain, arthralgia (joint pain) or swelling, enthesitis (inflammation of tendons and ligaments), and morning stiffness (2 questions: duration and severity). Each question is an easy to answer 10 centimeter (cm) visual analog scale (VAS), with 0 being none, and 10 being very severe. In order to give each of the 5 symptoms equal weight, the mean of the 2 questions about morning stiffness will be added to the total of the remaining 4 scores, and the final BASDAI score (ranging 0-10) is the average of the overall total score. Higher BASDAI score indicates more severe AS symptom.
Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score at Week 28 | Baseline and Week 28
  The BASDAI is used to measure the ankylosing spondylitis (AS) disease severity. It consists of 6 questions: fatigue, spinal pain, arthralgia (joint pain) or swelling, enthesitis (inflammation of tendons and ligaments), and morning stiffness (2 questions: duration and severity). Each question is an easy to answer 10cm visual analog scale (VAS), with 0 being none, and 10 being very severe. In order to give each of the 5 symptoms equal weight, the mean of the 2 questions about morning stiffness will be added to the total of the remaining 4 scores, and the final BASDAI score (ranging 0-10) is the average of the overall total score. Higher BASDAI score indicates more severe AS symptom.
Treatment Retention | Time from first ustekinumab administration to drug stop or switch or study withdrawal (approximately up to 28 weeks)
  Time from first ustekinumab administration to drug stop or switch or study withdrawal will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Cilag S.A.S., France Clinical Trial, Study Director — Janssen Cilag S.A.S.
Locations (1):
- Hôpital Edouard Herriot, Lyon, France